CLINICAL TRIAL: NCT01918865
Title: A Double Blind, Placebo-Controlled, Phase 2 Study to Assess the Safety, Tolerability, and Efficacy of ISIS 404173 Administered Once Weekly to Obese Patients With Type 2 Diabetes Mellitus Being Treated With Metformin or Metformin Plus Sulfonylurea
Brief Title: Safety, Tolerability, and Efficacy of ISIS-PTP1BRx in Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ISIS 404173-CS2
Record Dates: First submitted 2013-08-05; First posted 2013-08-08 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2014-09

CONDITIONS: Type 2 Diabetes Mellitus; Obese
Keywords: Type 2 Diabetes Mellitus; T2DM
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ISIS-PTP1BRx (Experimental): Weekly Dosing for 26 Weeks
  Interventions: Drug: ISIS-PTP1BRx; Drug: daily OAD (metformin and/or sulfonylurea)
- Placebo (Placebo Comparator): Weekly Dosing for 26 Weeks
  Interventions: Drug: Placebo; Drug: daily OAD (metformin and/or sulfonylurea)

INTERVENTIONS:
Drug: ISIS-PTP1BRx
  Arms: ISIS-PTP1BRx
Drug: Placebo
  Arms: Placebo
Drug: daily OAD (metformin and/or sulfonylurea)

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and efficacy of ISIS-PTP1BRx + oral antidiabetic drug/s (metformin and/or sulfonylurea) versus placebo + oral antidiabetic drug/s.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) >/= 27 kg/m2
* HbA1c between 7.5% and 10.5% (inclusive)
* C-Peptide (fasting) greater than or equal to 500 pmol/L
* On stable dose of metformin alone or in combination with a stable dose of sulfonylurea for >/= 3 months prior to screening, and remain on stable dose throughout the study
* Agree to conduct home-based (fasted) blood glucose testing as directed

Exclusion Criteria:

* Clinically significant abnormalities in medical history or physical exam
* Serum creatinine > ULN at Screening
* Clinical signs or symptoms of liver disease, acute or chronic hepatitis, or ALT or AST > 1.5x ULN at Screening
* History of renal transplantation or renal dialysis
* GFR < 60 mL/min at Screening
* History of diabetic ketoacidosis
* History of greater than 3 episodes of severe hypoglycemia within 6 months of screening
* Allergy to sulfur containing drugs
* Treatment with other drugs or medications not allowed per study specific Disallowed Concomitant Medicines
* Any other significant illness or condition that may interfere with the patient participating or completing the study
* Inability or unwillingness to comply with protocol or study procedures

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2013-08; Primary Completion 2014-10 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Incidence, severity, dose-relationship of adverse effects, and changes in laboratory evaluations as a measure of safety | 38 weeks
Change in plasma HbA1c levels at Week 27 compared to Baseline as a measure of efficacy | 27 weeks

SECONDARY OUTCOMES:
Change in FPG, weekly average SMPG, seven-point glucose profile, lipid profile, body weight, & BMI at Week 27 compared to Baseline as a measure of efficacy | 27 Weeks

CONTACTS AND LOCATIONS:
Locations (20):
- Argentina (2):
  - Isis Investigative Site, Mar del Plata, Buenos Aires
  - Isis Investigative Site, Rosario, Santa Fe Province
- Canada (7):
  - Isis Investigational Site, Edmonton, Alberta
  - Isis Investigational Site, Kelowna, British Columbia
  - Isis Investigational Site, Vancouver, British Columbia
  - Isis Investigational Site, Etobicoke, Ontario
  - Isis Investigational Site, Toronto, Ontario
  - Isis Investigative Site, Toronto, Ontario
  - Isis Investigational Site, Saskatoon, Saskatchewan
- South Africa (11):
  - Isis Investigational Site, Benoni, Benoni
  - Isis Investigational Site, Bloemfontein, Bloemfontein
  - Isis Investigational Site, Centurion, Gauteng
  - Isis Investigational Site, Mamelodi, Gauteng
  - Isis Investigational Site, Pretoria, Gauteng
  - Isis Investigational Site, Port Elizabeth, Korsten
  - Isis Investigational Site, Durban, KwaZulu-Natal
  - Isis Investigational Site, Middelburg, Mpumalanga
  - Isis Investigational Site, Pretoria, Pretoria
  - Isis Investigational Site, Limpopo, Thabazimbi
  - Isis Investigational Site, Cape Town, Western Cape

REFERENCES:
- [Derived] Digenio A, Pham NC, Watts LM, Morgan ES, Jung SW, Baker BF, Geary RS, Bhanot S. Antisense Inhibition of Protein Tyrosine Phosphatase 1B With IONIS-PTP-1BRx Improves Insulin Sensitivity and Reduces Weight in Overweight Patients With Type 2 Diabetes. Diabetes Care. 2018 Apr;41(4):807-814. doi: 10.2337/dc17-2132. Epub 2018 Feb 9. PMID 29439147